CLINICAL TRIAL: NCT04180956
Title: Reducing Racial Disparities in Healthcare: Developing Social Connections Through Behavioral Science
Brief Title: Addressing Microaggressions in Racially Charged Patient-provider Interactions: A Pilot Randomized Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Bastyr University (Other)
Responsible Party: Principal Investigator, Jonathan Kanter, Research Associate Professor, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: Bastyr_16-1557
Record Dates: First submitted 2018-10-30; First posted 2019-11-29 (Actual); Last update posted 2019-12-03 (Actual); Status verified 2019-11

CONDITIONS: Racism
MeSH Terms: conditions — Racism

STUDY DESIGN:
Intervention Model Description: This is a randomized controlled trial, wherein doctors are prospectively assigned to either an intervention or waitlist control condition.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The participants, who are the care providers, are blind to condition in that they are simply told when to show up for patient exams and the workshop (intervention condition). The outcomes assessors who rated microaggressions was blind to condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The bias-reduction intervention opened with a didactic on health disparities, stereotypes, microaggressions, interracial provider-patient interactions and racism. Then, a guided, interracial eye-contact mindfulness exercise was performed to increase providers' awareness and acceptance of subtle bias that occurs in interracial interactions. Then, in small, mixed-race groups, participants practiced the above mindfulness skills while reciprocally sharing and responding with empathy to each other's personal life histories and personal narratives of loss and/or betrayal. The intervention ended with explicit practice component, involving practice and feedback.
  Interventions: Other: Bias-reduction Intervention
- Control (No Intervention): The control condition was a waitlist condition. Doctors were given workshop materials after the study ended.

INTERVENTIONS:
Other: Bias-reduction Intervention — A training for doctors
  Arms: Intervention

SUMMARY:
Racial bias in medical care is a significant public health issue, with increased focus on microaggressions and the quality of patient-provider interactions. Innovations in training interventions are needed to decrease microaggressions and improve provider communication and rapport with patients of color during medical encounters. This paper presents a pilot randomized trial of an innovative clinical workshop that employed a theoretical model from social and contextual behavioral sciences. The intervention was largely informed by research on the importance of mindfulness and interracial contact involving reciprocal exchanges of vulnerability and responsiveness, to target processes centered on the providers' likelihood of expressing biases and negative stereotypes when interacting with patients of color in racially challenging moments. Twenty-five medical student and recent graduate participants were randomized to a workshop intervention or no intervention. Outcomes were measured via provider self-report and observed changes in targeted provider behaviors. Specifically, two independent, blind teams of coders assessed provider emotional rapport and responsiveness during simulated interracial patient encounters with standardized Black patients who presented specific racial challenges to participants. We observed greater improvements in observed emotional rapport and responsiveness (indexing fewer microaggressions), improved self-reported explicit attitudes toward minoritized groups, and improved self-reported working alliance and closeness with the Black standardized patients were observed and reported by intervention participants. Effects largely were driven by improvements by the White participants.

ELIGIBILITY:
Inclusion Criteria:

* Medical students or recent graduates of Bastyr University.

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2016-05-24 (Actual); Primary Completion 2016-09-25 (Actual); Study Completion 2016-09-25 (Actual)

PRIMARY OUTCOMES:
Change in Emotional Rapport Building from Pre- to Post-Intervention | Pre-test occurred on Day 1, the Intervention occurred Day 2, and then post-test occurred Day 4ater after the intervention
  We used the Roter Interactional Analysis System (RIAS), a turn-by-turn coding system in which each provider and patient utterance is coded into one of 40 categories of speech, which can be combined to create various summary scores. RIAS codes have demonstrated validity with a variety of samples and medical contexts. For the current study, two trained RIAS coders provided ratings, and both coders coded a subset of tapes (10%) for reliability (r= 0.92). Because standardized patients in our study were following a protocol and not responding naturally, we analyzed only provider codes, specifically the Emotional Rapport Building summary score which is a composite of doctor codes including emotional statements, legitimizing statements, concern statements, partnership statements, self-disclosure statements, and reassurance statements.
Change in responsiveness to racial challenges from Pre- to Post-Intervention | Pre-test occurred on Day 1, the Intervention occurred Day 2, and then post-test occurred Day 4ater after the intervention
  We modified observer-based responsiveness coding systems used in previous research that operationalized positive responsiveness in dyads as concrete instances of understanding, validation, and caring on a 0 to 3 scale. We expanded the previous 0 code, which originally combined both no responses (e.g., simply ignoring the challenge) and invalidating responses (e.g., defensive or microaggressive responses), into a negative responsiveness dimension and provided anchors and examples for each score, producing a Likert scale from - 3 to + 3, as shown in Table 3. Four coders were trained to high reliability.

SECONDARY OUTCOMES:
Change in offensiveness from Pre- to Post-Intervention | Pre-test occurred on Day 1, the Intervention occurred Day 2, and then post-test occurred Day 4
  Single-item question analyzed by responsiveness coders, asking "did the doctor say anything offensive?"
Change in Bias from Pre- to Post-Intervention | Pre-test occurred on Day 1, the Intervention occurred Day 2, and then post-test occurred Day 4
  Single-item question analyzed by responsiveness coders, asking "Was the doctor overtly biased against the patient?"
Change in Recommendations from Pre- to Post-Intervention | Pre-test occurred on Day 1, the Intervention occurred Day 2, and then post-test occurred Day 4
  Single-item question analyzed by responsiveness coders, asking "Would you recommend that a Black friend with the same problem as this patient see this doctor over any other doctor?"
Change in Patient experience from Pre- to Post-Intervention | Pre-test occurred on Day 1, the Intervention occurred Day 2, and then post-test occurred Day 4
  Single-item question analyzed by responsiveness coders, asking "Do you think the patient had a positive experience?"
Change in Ethnocultural empathy from Pre- to Post-Intervention | Pre-test occurred on Day 1, the Intervention occurred Day 2, and then post-test occurred Day 4
  Everyday Multicultural Competencies/Revised Scale of Ethnocultural Empathy (EMC/RSEE), which has strong evidence for factor structure, reliability and discriminant validity. There are multiple subscales; we were interested in empathic perspective-taking and acting as an ally
Change in attitudes toward various ethnic/racial groups from Pre- to Post-Intervention | Pre-test occurred during screening, between 5 days and 4 months prior to Intervention; post-test occurred two days after intervention.
  To assess explicit attitudes towards various ethnic and racial groups, participants provided feeling thermometer ratings for different groups of people, including African Americans and 13 other demographic categories, from 0 (extremely unfavorable) to 100 (extremely favorable). Low scores on feeling thermometers are interpreted as a simple indicator of explicit prejudice.
Change in Working alliance from Pre- to Post-Intervention | Pre-test occurred on Day 1, the Intervention occurred Day 2, and then post-test occurred Day 4
  After each standardized patient interaction, participants completed the 12-item Bond subscale of the Working Alliance Inventory (WAI), a widely used measure to assess the provider-patient alliance in therapeutic interactions. Bond subscale items ask about specific feelings toward the patient, including "I respect this patient."
Change in Interaction closeness from Pre- to Post-Intervention | Pre-test occurred on Day 1, the Intervention occurred Day 2, and then post-test occurred Day 4
  After each standardized patient interaction, participants answered three questions about their experience of the interaction. First, they completed the Inclusion of the Other in the Self (IOS) scale, a well-validated, single-item, pictorial measure of relational closeness which has been used to assess closeness in interracial contexts and between patients and providers. The other two closeness items were the following: 1) Relative to all your other relationships with patients (outside of this study), how would you characterize your relationship with this patient? and 2) Relative to what you know about other patient's relationships with their doctors, how would you characterize your relationship with this patient? Agreement with these items was assessed on a 7-point Likert scale ranging from 1 (less close) to 7 (more close).

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Kanter, Ph.D., Principal Investigator — University of Washington
Locations (1):
- Bastyr University Seattle Clinic, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No
IPD will be shared by request so as not to violate individual privacy concerns.